CLINICAL TRIAL: NCT02885090
Title: Search for New Genes Involved in Molecular Etiology of Rett Syndrome Through Comparative Genomic Hybridization on DNA Microarrays
Brief Title: New Genes Involved in Molecular Etiology of Rett Syndrome Through DNA Microarray Comparative Genomic Hybridization
Acronym: RETT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-A01147-50
Record Dates: First submitted 2016-08-23; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RTT patient (Experimental): Blood sampling
  Interventions: Procedure: Blood sampling
- Parents (Experimental): Blood sampling. To distinguish between inherited polymorphic variants and potentially deleterious new imbalances.
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — In children: 2 EDTA tubes of 7 ml, 1 Heparin Li tube of 5 ml and 2 PAXgene tubes of 2.5 ml (max 0.8-0.9 ml blood/kg) In parents: 2 EDTA tubes of 7 ml, 1 Heparin Li tube of 5 ml.

SUMMARY:
Rett syndrome (RTT) is a genetic encephalopathy and the typical form is caused by mutations in the gene MECP2. It is a genetically heterogeneous pathology. CDKL5 and FOXG1 have been recently discovered being involved in other forms of RTT. However, at least 5% of typical forms and more other atypical forms are not linked to any of 3 genes known to be involved in the disease.

The purpose of this study is to identify new genes involved in molecular etiology of typical and atypical forms of RTT.

DETAILED DESCRIPTION:
Search for pathogenic chromosomal imbalance through comparative genomic hybridization (aCGH) on DNA microarrays will be done in a group of patients having typical or atypical forms of RTT without known mutations in MECP2, CDKL5 et FOXG1B genes.

After imbalance confirmation by qPCR, the pathogenic potential of the segmental aneusomy will be assigned according to the interpretation of aCGH technique-dedicated DECEPHER, BACH and GVD databases. Analysis of parents will allow distinguishing between inherited polymorphic variants and potentially deleterious new imbalances.

In case of a new imbalance, a bioinformatics approach will look for candidate genes that will be possibly confirmed by classic mutation screening (sequencing and PCR) in all typical and atypical cases of RTT present in the cohort.

The identification of new genes involved in RTT will ameliorate the molecular diagnosis of the disease and genetic counseling for families. This project will allow progression in comprehension of physiopathological mechanisms of cerebral development abnormalities

ELIGIBILITY:
Inclusion Criteria:

* Patients: RETT syndrome
* Patients: Female
* Parents: parent of a patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Analysis of chromosomal imbalances through comparative genomic hybridization on DNA microarrays | up to 12 months
  Search for pathogenic chromosomal imbalance

CONTACTS AND LOCATIONS:
Overall Officials: Christophe PHILIPPE,, Principal Investigator — Laboratoire de Génétique Médicale, Rue du Morvan, 54511 Vandoeuvre-Les-Nancy Cédex
Locations (9):
- France (9):
  - Handicaps de l'Enfant - Pavillon Ste Marie, CHU St Jacques, Besançon
  - Service de Neuropédiatrie, Hôpital St Jacques, CHU de Besançon, Besançon
  - Unité de génétique, Groupe hospitalier Hôpital Flaubert, Caen
  - Centre de Génétique Hôpital d'Enfants, CHU de Dijon, Dijon
  - Service de neuropédiatrie, CHU Hôpital Gui de Chauliac, Montpellier
  - Laboratoire de Génétique chromosomique, CHU Hôpital l'Archet 2, Nice
  - Service de génétique médicale, CHU Hôpital Purpan, Nice
  - Service de génétique médicale, CHU Hôpital Purpan, CHU de Toulouse, Toulouse
  - Laboratoire de Génétique, Hôpitaux de Brabois, CHU de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No